CLINICAL TRIAL: NCT04712019
Title: A Randomized Controlled Trial Evaluating Edema and ROM Using Negative Pressure Therapy Over Closed Incisions and Surrounding Soft Tissue Versus Standard Surgical Dressings in Bilateral Total Knee Arthroplasty: A Pilot Study
Brief Title: Evaluating Edema and Range of Motion Using Negative Pressure Therapy vs. Standard Surgical Dressing in Bilateral TKA
Acronym: ENABLE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREVENA.RESTOR.ARTHRO.2019.01
Record Dates: First submitted 2021-01-14; First posted 2021-01-15 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Surgical Wound; Bilateral Total Knee Arthroplasty; Wounds and Injuries; Joint Diseases; Musculoskeletal Diseases; Edema Leg; Joint Pain; Arthritis Knee
MeSH Terms: conditions — Surgical Wound; Wounds and Injuries; Joint Diseases; Musculoskeletal Diseases; Arthralgia

STUDY DESIGN:
Intervention Model Description: One leg receives ciNPT and the other leg receives standard silver containing dressing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Closed Incision Negative Pressure Therapy (ciNPT) Dressing (Experimental): Prevena Restor Arthro-Form Dressing with Prevena Plus Therapy Unit
  Interventions: Device: Closed Incision Negative Pressure Therapy (ciNPT)
- Standard Silver-containing Dressing (Active Comparator): Standard silver dressing - standard of care at hospital
  Interventions: Device: Standard Silver-containing Dressing

INTERVENTIONS:
Device: Closed Incision Negative Pressure Therapy (ciNPT) — Closed Incision Negative Pressure Therapy applied through a foam bolster with a wicking interface fabric at 125mmHg of continuous negative pressure on a closed surgical incision
  Other Names: Prevena Restor ArthroForm; Prevena Plus 125 Therapy Unit
  Arms: Closed Incision Negative Pressure Therapy (ciNPT) Dressing
Device: Standard Silver-containing Dressing — A standard silver-containing dressing applied to a closed surgical incision
  Arms: Standard Silver-containing Dressing

SUMMARY:
This study will compare the effects of closed incision negative pressure dressing vs. standard of care silver dressing on lower limb swelling after bilateral primary total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* is at least 22 years of age on the date of informed consent.
* can independently provide informed consent.
* requires and is scheduled to undergo a simultaneous, bilateral, primary TKA.
* is willing and physically capable of undergoing a simultaneous, bilateral, primary TKA with or without replacement of the patella.
* is willing and able to return for all scheduled study visits.

Exclusion Criteria:

* is pregnant or lactating.
* has signs of an infection in the area of either knee or has signs of a systemic infection at the time of surgery.
* is a chronic opioid user, defined per the CDC guidelines as opioid use for >3 months, at the time of enrollment.
* has a current diagnosis of lymphedema in either leg.
* has signs, symptoms, or a current diagnosis of venous insufficiency in either leg, as determined by the investigator's review of the subject's medical history.
* has a history of clotting disorder or prior history of deep vein thrombosis
* will undergo a unilateral TKA.
* will undergo a staged, bilateral TKA.
* has had previous knee replacement surgery.
* has received a corticosteroid injection into either knee within 30 days of surgery.
* undergoes a simultaneous, bilateral TKA with a planned different incision type on each knee (eg, midline incision vs. medial parapatellar incision).
* has known sensitivity to the study product components (drape and/or dressing materials in direct contact with the closed incision or skin).
* has known sensitivity to silver.
* is enrolled in another interventional clinical study.
* has skin cancer localized at or in proximity to the incision site.
* does not have access to an electronic device (smartphone, iPad, or computer) on a daily basis to complete online assessments.
* has condition(s) that, in the opinion of the investigator, cause the subject to be an overall health risk that is unsuitable for the surgery.
* has condition(s) that, in the opinion of the investigator, will impact study endpoints (eg, hemophilia or autoimmune disorders) or the ability to comply with study procedures.

Intra-Op Exclusion Criteria:

* does not receive a "total" knee replacement for first knee. For example, a partial or uni-compartmental knee replacement is performed
* has a surgical incision that would preclude placement of either dressing onto the knee
* has a TKA resulting in a muscle flap

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Cushner, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (6):
- United States (6):
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Rubin Institute for Advanced Orthopedics, Baltimore, Maryland
  - Johns Hopkins Orthopaedics, Columbia, Maryland
  - Northwell Health - Southside Hospital, Bay Shore, New York
  - Northwell Health - Lenox Hill Hospital, New York, New York
  - Northwell Health - Long Island Jewish Valley Stream, Valley Stream, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of subjects enrolled is 10; however, each leg is a separate arm in the study allowing for a total of 20 treatment allocations. The number started will be 20 which is greater than the protocol enrollment wherever this is acceptable for paired study design.
Units Other Than Participants: Knee
Period: Overall Study
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Started | 10; 10 Knee | 10; 10 Knee
Completed | 7; 7 Knee | 7; 7 Knee
Not Completed | 3; 3 Knee | 3; 3 Knee
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol required withdrawal - crossover treatment | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Subjects - Both Arms: This study was a split subject design. All subjects received both treatments - one on each knee.
Arm/Group | All Enrolled Subjects - Both Arms
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
BMI [Mean (Standard Deviation); unit: kg/m2] | 31.8 (6.57)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Lower Limb Volume
Description: Percent change in lower limb volume as calculated using manual circumference measurements
Time Frame: 5-7 days after bilateral TKA procedure
Population: This is the full analysis set which excludes one subject who lacks data at the 5-7 day visit.
Measure: Mean (Standard Deviation); unit: percentage of change in lower leg volume
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 9 | 9
percentage of change in lower leg volume | 14.7 (15.48) | 13.3 (12.43)

2. Secondary Outcome: Percent Change in Lower Limb Volume
Description: Percent change in lower limb volume as calculated using manual circumference measurements
Time Frame: 12-14 days after bilateral TKA procedure
Population: This is the full analysis set which excludes two subjects who lack data at the 12-14 day visit.
Measure: Mean (Standard Deviation); unit: percentage of change in lower leg volume
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 8 | 8
percentage of change in lower leg volume | 16.0 (9.82) | 10.7 (21.88)

3. Secondary Outcome: Percent Change in Lower Limb Volume
Description: Percent change in lower limb volume as calculated using manual circumference measurements
Time Frame: 35-49 days after bilateral TKA procedure
Population: This is the full analysis set which excludes three subjects who lack data at the 35-49 day visit.
Measure: Mean (Standard Deviation); unit: percentage of change in lower leg volume
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 7 | 7
percentage of change in lower leg volume | 1.4 (6.40) | 1.6 (6.12)

4. Secondary Outcome: Percent Change in Lower Limb Volume
Description: Percent change in lower limb volume as calculated using manual circumference measurements
Time Frame: 77-91 days after bilateral TKA procedure
Population: This is the full analysis set which excludes three subjects who lack data at the 77-91 day visit.
Measure: Mean (Standard Deviation); unit: percentage of change in lower leg volume
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 7 | 7
percentage of change in lower leg volume | -1.3 (9.58) | -4.4 (6.51)

5. Secondary Outcome: Percent Change in Lower Limb Circumference
Description: Percent change in circumferences measured at 10 cm above the center of the patella, at the center of patella and 10cm below the center of the patella
Time Frame: 5-7 days after bilateral TKA procedure
Population: This is the full analysis set which excludes one subject who lacks data at the 5-7 day visit.
Measure: Mean (Standard Deviation); unit: % change in lower leg circumference
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 9 | 9
% change in lower leg circumference
  10cm above Patella | 13.2 (5.84) | 7.8 (6.75)
  Center of Patella | 7.7 (11.23) | 6.4 (7.89)
  10cm below Patella | 3.6 (5.28) | 5.3 (5.06)
  at the ankle, 1cm above medial malleolus | NA (NA) — Collected values were below the lower limit of qualification | NA (NA) — Collected values were below the lower limit of qualification

6. Secondary Outcome: Percent Change in Lower Limb Circumference
Description: as for outcome 5
Time Frame: 12-14 days after bilateral TKA procedure
Population: This is the full analysis set which excludes two subjects who lack data at the 12-14 day visit.
Measure: Mean (Standard Deviation); unit: % change in lower leg circumference
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 8 | 8
% change in lower leg circumference
  10cm above Patella | 8.4 (4.37) | 9.8 (5.42)
  Center of Patella | 12.8 (5.03) | 2.2 (25.01)
  10cm below Patella | 3.9 (7.44) | 3.6 (9.14)
  at the ankle, 1cm above medial malleolus | NA (NA) — Collected values were below the lower limit of qualification | NA (NA) — Collected values were below the lower limit of qualification

7. Secondary Outcome: Percent Change in Lower Limb Circumference
Description: as for outcome 5
Time Frame: 35-49 days after bilateral TKA procedure
Population: This is the full analysis set which excludes three subjects who lack data at the 35-49 day visit.
Measure: Mean (Standard Deviation); unit: % change in lower leg circumference
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 7 | 7
% change in lower leg circumference
  10cm above Patella | 2.0 (3.04) | 0.7 (4.93)
  Center of Patella | 1.9 (4.24) | 3.0 (3.15)
  10cm below Patella | 0.0 (5.20) | -0.9 (5.96)
  at the ankle, 1cm above medial malleolus | NA (NA) — Collected values were below the lower limit of qualification | NA (NA) — Collected values were below the lower limit of qualification

8. Secondary Outcome: Percent Change in Lower Limb Circumference
Description: as for outcome 5
Time Frame: 77-91 days after bilateral TKA procedure
Population: This is the full analysis set which excludes three subjects who lack data at the 77-91 day visit.
Measure: Mean (Standard Deviation); unit: % change in lower leg circumference
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 7 | 7
% change in lower leg circumference
  10cm above Patella | 0.1 (5.38) | -3.6 (5.41)
  Center of Patella | -0.5 (5.04) | -0.3 (2.65)
  10cm below Patella | -0.9 (7.44) | -3.8 (7.08)
  at the ankle, 1cm above medial malleolus | NA (NA) — Collected values were below the lower limit of qualification | NA (NA) — Collected values were below the lower limit of qualification

9. Secondary Outcome: Change in Knee Flexion Angle
Description: Change in knee flexion angle from baseline to Visit 3
Time Frame: 5-7 days after bilateral TKA procedure
Population: This is the full analysis set which excludes three subjects who lack data at the 5-7 day visit.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 7 | 7
Degrees | -18.3 (22.02) | -19.9 (17.39)

10. Secondary Outcome: Change in Knee Flexion Angle
Description: Change in knee flexion angle from baseline to Visit 4
Time Frame: 12-14 days after bilateral TKA procedure
Population: This is the full analysis set which excludes three subjects who lack data at the 12-14 day visit.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 7 | 7
Degrees | -10.7 (25.36) | -9.6 (18.65)

11. Secondary Outcome: Change in Knee Flexion Angle
Description: Change in knee flexion angle from baseline to Visit 5
Time Frame: 35-49 days after bilateral TKA procedure
Population: This is the full analysis set which excludes three subjects who lack data at the 35-49 day visit.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 7 | 7
Degrees | 0.0 (21.98) | 1.0 (11.42)

12. Secondary Outcome: Change in Knee Flexion Angle
Description: Change in knee flexion angle from baseline to Visit 6
Time Frame: 77-91 days after bilateral TKA procedure
Population: This is the full analysis set which excludes three subjects who lack data at the 77-91 day visit.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 7 | 7
Degrees | 17.9 (22.52) | 15.7 (13.97)

13. Secondary Outcome: Change in Knee Extension Angle
Description: Change in knee extension angle from baseline to Visit 3
Time Frame: 5-7 days after bilateral TKA procedure
Population: This is the full analysis set which excludes three subjects who lack data at the 5-7 day visit.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 7 | 7
Degrees | -2.9 (4.10) | 1.1 (7.97)

14. Secondary Outcome: Change in Knee Extension Angle
Description: Change in knee extension angle from baseline to Visit 4
Time Frame: 12-14 days after bilateral TKA procedure
Population: This is the full analysis set which excludes three subjects who lack data at the 12-14 day visit.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 7 | 7
Degrees | 9.0 (26.95) | 2.3 (6.24)

15. Secondary Outcome: Change in Knee Extension Angle
Description: Change in knee extension angle from baseline to Visit 5
Time Frame: 35-49 days after bilateral TKA procedure
Population: This is the full analysis set which excludes three subjects who lack data at the 35-49 day visit.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 7 | 7
Degrees | -2.4 (3.36) | 1.6 (6.40)

16. Secondary Outcome: Change in Knee Extension Angle
Description: Change in knee extension angle from baseline to Visit 6
Time Frame: 77-91 days after bilateral TKA procedure
Population: This is the full analysis set which excludes three subjects who lack data at the 77-91 day visit.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 7 | 7
Degrees | -2.9 (7.76) | 0.3 (9.25)

17. Secondary Outcome: Change of Total Range of Motion in Degrees
Description: Change of total ROM degrees, defined as the flexion angle minus the extension angle from baseline to Visit 3
Time Frame: 5-7 days after bilateral TKA procedure
Population: This is the full analysis set which excludes three subjects who lack data at the 5-7 day visit.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 7 | 7
Degrees | -15.4 (23.19) | -21.0 (20.12)

18. Secondary Outcome: Change of Total Range of Motion in Degrees
Description: Change of total ROM degrees, defined as the flexion angle minus the extension angle from baseline to Visit 4
Time Frame: 12-14 days after bilateral TKA procedure
Population: This is the full analysis set which excludes three subjects who lack data at the 12-14 day visit.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 7 | 7
Degrees | -19.7 (49.54) | -11.9 (21.80)

19. Secondary Outcome: Change of Total Range of Motion in Degrees
Description: Change of total ROM degrees, defined as the flexion angle minus the extension angle from baseline to Visit 5
Time Frame: 35-49 days after bilateral TKA procedure
Population: This is the full analysis set which excludes three subjects who lack data at the 35-49 day visit.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 7 | 7
Degrees | 2.4 (24.96) | -0.6 (12.43)

20. Secondary Outcome: Change of Total Range of Motion in Degrees
Description: Change of total ROM degrees, defined as the flexion angle minus the extension angle from baseline to Visit 6
Time Frame: 77-91 days after bilateral TKA procedure
Population: This is the full analysis set which excludes three subjects who lack data at the 77-91 day visit.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 7 | 7
Degrees | 20.7 (28.40) | 15.4 (19.01)

21. Secondary Outcome: Incidence of Surgical Site Complications (SSCs)
Description: Incidence of surgical site complications defined as:
  * Superficial Surgical Site Infection (SSI)
  * Deep SSI
  * Full thickness skin dehiscence
  * Seroma or hematoma requiring drainage or surgery
  * Skin necrosis
  * Continued drainage at the time of dressing removal
Time Frame: within 49 days of bilateral TKA procedure
Population: This is the full analysis set which excludes three subjects who lack data as of Day 49.
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 7 | 7
Participants | 0 | 0

22. Secondary Outcome: Incidence of Surgical Site Complications (SSCs)
Description: as for outcome 21
Time Frame: within 91 days of bilateral TKA procedure
Population: This is the full analysis set which excludes three subjects who lack data as of Day 91.
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 7 | 7
Participants | 0 | 0

23. Secondary Outcome: Scar Cosmesis Assessment
Description: Validated tool to assess the quality of postoperative scars in clinical and research settings. Scores range from 4 (best) to 14 (worst). Due to the lack of subjects and study data, only the value recorded at the final study visit was analyzed for each subject. The average score for each study arm was then calculated with the available data.
Time Frame: Long Term Follow-up occurring 77-91 days after bilateral TKA procedure
Population: This is the full analysis set which excludes three subjects who did not complete study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 7 | 7
units on a scale | 5.86 (1.069) | 6.43 (1.902)

24. Secondary Outcome: Average Pain in Each Leg in the Last 24 Hours
Description: The average pain in each leg in the last 24 hours, using an NPRS (numerical pain rating scale) of 0-10. 0 represents No Pain with 10 representing Extremely Painful. Due to the lack of subjects and study data, only the last recorded pain value was analyzed for each subject. The average score for each study arm was then calculated with the available data.
Time Frame: End of Treatment Visit occurring 12-14 days after bilateral TKA procedure
Population: This is the full analysis set of available data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 2 | 2
score on a scale | 5.00 (4.243) | 5.00 (4.243)

25. Secondary Outcome: Worst Pain in Each Leg in the Last 24 Hours
Description: The worst pain in each leg in the last 24 hours, using an NPRS of 0-10. 0 represents No Pain with 10 representing Extremely Painful. Due to the lack of subjects and study data, only the last recorded pain value was analyzed for each subject. The average score for each study arm was then calculated with the available data.
Time Frame: End of Treatment Visit occurring 12-14 days after bilateral TKA procedure
Population: This is the full analysis set of available data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) Dressing | Standard Silver-containing Dressing
Number analyzed (Participants) | 2 | 2
score on a scale | 6.00 (4.243) | 5.50 (4.950)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of randomization through completion of the Visit 6 (77-91 days Post-op)
Groups:
- All Enrolled Subjects - Both Arms: Subjects who received both the Prevena Restor Arthro-Form Dressing with Prevena Plus Therapy Unit and Standard Silver-containing Dressing: A standard silver-containing dressing applied to a closed surgical incision.
Arm/Group | All Enrolled Subjects - Both Arms
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects - Both Arms (N=10)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects - Both Arms (N=10)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) — This adverse event of blister affected the ciNPT arm and related to treatment.
Hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination of the study due to inability to enroll in the trial lead to a small number of subjects analyzed as well as incomplete data assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT04712019/Prot_SAP_000.pdf